CLINICAL TRIAL: NCT03540784
Title: Effect of Whole-body Electromyostimulation Combined With a High Protein Diet in Malnourished Patients With Inflammatory Bowel Disease
Brief Title: Effects of WB-EMS and High Protein Diet in IBD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CED EMS
Record Dates: First submitted 2018-05-15; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Inflammatory Bowel Diseases
Keywords: muscle weakness; muscle mass; whole-body electromyostimulation; WB-EMS; nutrition; protein; crohn's disease; ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Muscle Weakness; Crohn Disease; Colitis, Ulcerative | interventions — Nutritional Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): usual care treatment
- Nutrition (Experimental): high-protein nutrition therapy
  Interventions: Other: Nutritional support
- EMS+Nutrition (Experimental): WB-EMS Training (2x/week á 20 min) + high-protein nutrition therapy
  Interventions: Other: WB-EMS; Other: Nutritional support

INTERVENTIONS:
Other: WB-EMS — WB-EMS training is performed 2x/week for 12 weeks; Stimulation protocol: Frequency of 85 Hz, pulse duration of 0.35 ms, stimulation period of 6 sec, resting period of 4 sec; supervised by certified training instructors/physiotherapists participants perform simple exercises during the stimulation period following a video tutorial
  Arms: EMS+Nutrition
Other: Nutritional support — dietary monitoring by dietary records; nutritional counselling by dietician, dietary advices: 1.5 g/kg bodyweight/day
  Arms: EMS+Nutrition; Nutrition

SUMMARY:
Patients with inflammatory bowel disease (IBD) often suffer from muscle weakness and a low bone mineral density as a consequence of systemic Inflammation and disease treatment limiting Quality of life in a considerable way. Exercise interventions to build up muscle mass and increasing physical function are promising Tools to improve the whole muscular Status of those patients. However, in the acute Phase of IBDs conventional Training methods may be too strenous, also because patients are suffering from acute gastrointestinal symptoms and feel fatigued. Due to those symptoms, patients present low Food intake and great loss of nutrients and energy especially by diarrhea. Individualized nutritional Support may be helpful to avoid malnutrition. The aim of this pilot study is to investigate the effect of a combined exercise and Nutrition Intervention using the gentle Training method of whole-body electromyostimulation (WB-EMS) combined with a individual high Protein nutritional Support on muscle mass, Body composition, physical function, Quality of life and gastrointestinal symptoms in outpatients with IBD.

ELIGIBILITY:
Inclusion Criteria:

* outpatients with inflammatory bowel disease (Crohn's disease, ulcerative Colitis)
* adults (18 years and older)

Exclusion Criteria:

* simultaneous participation in other nutritional or exercise intervention Trials
* acute cardiovascular events
* use of anabolic medications
* epilepsy
* severe neurological diseases
* skin lesions in the area of electrodes
* energy active metals in body
* pregnancy
* acute vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2013-10-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle mass | 12 weeks
  assessed by bioelectrical impedance analysis in kg

SECONDARY OUTCOMES:
Body composition | 12 weeks
  assessed by bioelectrical impedance analysis in kg or %
Physical function - isometric muscle strength | 12 weeks
  isometric hand grip strength assessed by hand dynamometer
Physical function - Endurance | 12 weeks
  Six-minute-walk test (walking distance in m)
Physical function - lower limb strength | 12 weeks
  isometric lower limb strength assessed by isometric force plates in N
Quality of Life | 12 weeks
  IBDQ-D
Physical activity | 12 weeks
  IPAQ
Disease activity (Crohn's disease) | 12 weeks
  Harvey Bradshaw Index
Disease activity (ulcerative colitis) | 12 weeks
  Mayo Score
Inflammation status | 12 weeks
  C-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Erlangen, Medizinische Klinik 1, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No